CLINICAL TRIAL: NCT03096223
Title: A Phase 1, Open-Label, Multiple-Dose Study of KHK4083 in Subjects With Atopic Dermatitis
Brief Title: A Phase 1 Study of KHK4083 in Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4083-004
Record Dates: First submitted 2017-03-23; First posted 2017-03-30 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — KHK4083

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KHK4083 (Experimental)
  Interventions: Drug: KHK4083

INTERVENTIONS:
Drug: KHK4083 — IV administration

SUMMARY:
The objective of this study is to evaluate the safety and tolerability of multiple intravenous (IV) infusions of KHK4083 in subjects with moderate or severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent to participate in the study
2. Atopic dermatitis diagnosed according to the Definition and Diagnostic Criteria for Atopic Dermatitis (Guidelines for Management of Atopic Dermatitis 2016) established by the Japanese Dermatological Association
3. Moderate or severe (≥4.5) symptoms of atopic dermatitis at screening, according to the Rajka & Langeland Severity Index
4. Investigator Global Assessment(IGA) ≥3 (moderate) at screening

Exclusion Criteria:

1. Any of the following clinically significant concurrent illnesses:

   * Type 1 diabetes
   * Poorly controlled type 2 diabetes (HbA1c >8.5%)
   * Congestive heart failure (class II to IV of the New York Heart Association classification)
   * Myocardial infarction within 1 year
   * Unstable angina pectoris within 1 year
   * Poorly controlled hypertension (systolic pressure >150 mm Hg or diastolic pressure >90 mm Hg at screening)
   * Severe chronic lung diseases requiring oxygen therapy
   * Multiple sclerosis or other demyelinating diseases
   * Active malignancies, or onset or a history of treatment of malignancies within 5 years prior to informed consent (except for resected or surgically cured epithelial carcinoma of the uterine cervix, cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, or ductal carcinoma)
2. Current or past history of clinically significant cardiovascular, liver, renal, respiratory, hematologic, central nervous system, psychiatric, or autoimmune diseases/disorders other than those in 1)
3. Alcohol dependence, or drug dependence or a positive result for any of the drug abuse test items
4. Past or current history of drug allergy
5. Any clinically significant infection requiring hospitalization or IV administration of antibiotics within 8 weeks prior to pre-enrollment
6. Any planned surgical treatment during the study
7. Any skin disease that may affect the clinical symptom assessment
8. Pregnant or lactating women, or women willing to have a child during the study period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) or drug-related TEAEs and their nature | Up to 22 weeks post drug administration

SECONDARY OUTCOMES:
Serum KHK4083 concentration | Up to 22 weeks post drug administration
Maximum concentration (Cmax) | Up to 22 weeks post drug administration
Time to reach Cmax (tmax) | Up to 22 weeks post drug administration
Area under the curve (AUC) | Up to 22 weeks post drug administration
Anti-KHK4083 antibody production | Up to 22 weeks post drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Closed information, Sapporo, Japan

IPD SHARING:
Plan to Share IPD: Undecided